CLINICAL TRIAL: NCT01334268
Title: A Randomized Controlled Trial of the Resolute Zotarolimus-Eluting Stent Versus the Taxus Liberte Paclitaxel-Eluting Stent for Percutaneous Coronary Intervention in a Real-World All-comer Patient Population in China
Brief Title: RESOLUTE China RCT
Acronym: R-China RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IP 10009066DOC
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Ischemic Heart Disease; Stenotic Coronary Lesion; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease
Keywords: In-stent Late Lumen Loss (LLL); TARGET VESSEL FAILURE (TVF); MYOCARDIAL INFARCTION (MI); TARGET VESSEL REVASCULARIZATION (TVR); TARGET LESION REVASCULARIZATION (TLR); TARGET LESION FAILURE (TLF); STENT THROMBOSIS; RESTENOTIC LESION; PERCUTANEOUS CORONARY INTERVENTION (PCI); REAL-WORLD; THE RANDOMIZED CONTROLLED TRIAL
MeSH Terms: conditions — Myocardial Ischemia; Cardiovascular Diseases; Arteriosclerosis; Coronary Artery Disease; Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taxus Liberte Paclitaxel-Eluting Coronary Stent System (Active Comparator): Subjects will be randomized to be treated with Taxus Liberte Paclitaxel-Eluting Coronary Stent System by an interactive voice response system (IVRS).
  Interventions: Device: Taxus Liberte Paclitaxel-Eluting Coronary Stent System
- Medtronic Resolute (Zotarolimus-eluting stent) (Experimental): Subjects will be randomized to be treated with Medtronic Resolute (Zotarolimus-eluting stent) by an interactive voice response system (IVRS).
  Interventions: Device: Resolute Zotarolimus-Eluting Coronary Stent System

INTERVENTIONS:
Device: Taxus Liberte Paclitaxel-Eluting Coronary Stent System — Taxus Liberte Paclitaxel-Eluting Coronary Stent System Implantation
  Other Names: Taxus
  Arms: Taxus Liberte Paclitaxel-Eluting Coronary Stent System
Device: Resolute Zotarolimus-Eluting Coronary Stent System — Resolute Zotarolimus-Eluting Coronary Stent System Implantation
  Other Names: Resolute
  Arms: Medtronic Resolute (Zotarolimus-eluting stent)

SUMMARY:
The primary objective of this study is to evaluate the in-stent late lumen loss (LLL) at 9 months, defined as the difference between the post-procedure minimal lumen diameter (MLD) and the follow-up angiography MLD, of the Resolute Zotarolimus-Eluting Coronary Stent System compared to Taxus Liberte Paclitaxel-Eluting Coronary Stent System in a real-world all-comer patient population requiring stent implantation.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, two-arm, open-label study, designed to assess the non-inferiority of Resolute stent compared to Taxus Liberte stent in in-stent late lumen loss.

The primary objective of this study is to evaluate the in-stent late lumen loss (LLL) at 9 months, defined as the difference between the post-procedure minimal lumen diameter (MLD) and the follow-up angiography MLD, of the Resolute Zotarolimus-Eluting Coronary Stent System compared to Taxus Liberte Paclitaxel-Eluting Coronary Stent System in a real-world all-comer patient population requiring stent implantation.

This trial will be conducted at approximately 20 sites and will enroll up to 400 subjects, randomized to the Resolute stent and Taxus Liberte stent in a 1:1 ratio. Subjects will be randomized using an interactive voice response system (IVRS).

Due to the design characteristics of the devices, the study investigators and operators can not be blinded. However, the clinical event adjudication committee, consisting of cardiologists who are not participating in the study, will be blinded for the treatment arm of the subjects to avoid a potential bias in the adjudication process of events.

ELIGIBILITY:
Inclusion Criteria:

Patient must meet all of the following criteria to be eligible for treatment in the trial:

1. Age ≥ 18 years or minimum age as required by local regulations
2. The patient is an acceptable candidate for treatment with a drug-eluting stent in accordance with the applicable guidelines on percutaneous coronary interventions, the Instructions for Use of the Resolute stent and Taxus Liberte stent and the Declaration of Helsinki
3. The patient or legal representative has been informed of the nature of the trial and has consented to participate and authorized the collection and release of his/her medical information by signing a Patient Informed Consent Form
4. Intention to electively implant at least one Resolute stent or Taxus Liberte stent
5. The patient is willing and able to cooperate with study procedures and required follow up visits

Exclusion Criteria:

Patients will be excluded from the trial if any of the following criteria are met:

1. Known intolerance to aspirin, clopidogrel or ticlopidin, heparin, bivalirudin, cobalt, nickel, chromium, molybdenum, 316L stainless steel, polymer coatings (e.g. Biolinx), zotarolimus, paclitaxel, rapamycin, tacrolimus, everolimus, or any other analogue or derivative, or contrast media
2. Women with known pregnancy or who are lactating
3. High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
4. Currently participating in another trial that has not completed the primary endpoint or that clinically interferes with the current trial requirements
5. Planned surgery within 6 months of PCI unless dual anti-platelet therapy is maintained throughout the peri-surgical period
6. Previous enrollment in the Resolute China RCT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
in-stent late lumen loss (LLL) | 9 months
  in-stent late lumen loss (LLL), defined as the difference between the post-procedure minimal lumen diameter (MLD) and the follow-up angiography MLD.

SECONDARY OUTCOMES:
Device success | at the end of the index procedure or during hospital stay
  Definition 1: The attainment of <50% residual stenosis of the target lesion using only the assigned device.
  Definition 2: The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using the assigned device only. These measurements will be made by the independent angiographic core laboratory. If the core laboratory is unable to assess the % residual stenosis, the Investigator's assessment as recorded in the CRF will be used for the statistical analysis.
Death | 30d, 6m, 12m, 2yr, 3yr, 4yr, 5yr
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
Myocardial infarction | 30d, 6m, 12m, 2yr, 3yr, 4yr, 5yr
  All myocardial infarction data will be reported per Medtronic historical protocol definitions and according the Academic Research Consortium (ARC) definitions.
MACE composite endpoint | 30d, 6m, 12m, 2yr, 3yr, 4yr, 5yr
  Death, myocardial infarction (MI) (Q wave and non-Q wave), emergent coronary bypass surgery (CABG), or clinically-driven repeat target lesion revascularization by percutaneous or surgical methods.
Composite endpoint of (all cause) mortality, Myocardial Infarction (Q-wave and non Q-wave) or (any) revascularization | 30d, 6m, 12m, 2yr, 3yr, 4yr, 5yr
  Mortality, Myocardial Infarction (Q-wave and non Q wave) or (any) revascularization.
All revascularizations | 30d, 6m, 12m, 2yr, 3yr, 4yr, 5yr
  Target Legion Revascularization (TLR), Target Vessel Revascularization (TVR) and Non-TVR.
Target lesion failure (TLF) | 30d, 6m, 12m, 2yr, 3yr, 4yr, 5yr
  A composite endpoint of cardiac death, target vessel myocardial infarction (Q wave and non Q wave) or clinically-driven target lesion revascularization (TLR) by percutaneous or surgical methods.
Target vessel failure (TVF) | 30d, 6m, 12m, 2yr, 3yr, 4yr, 5yr
  A composite endpoint of cardiac death, target vessel myocardial infarction, or clinically-driven target vessel revascularization(TVR.
Stent thrombosis | 30d, 6m, 12m, 2yr, 3yr, 4yr, 5yr
  As determined by Medtronic historic and ARC definitions.
Lesion success | At the end of the index procedure or during hospital stay
  Definition 1: The attainment of <50% residual stenosis of the target lesion using any percutaneous method.
  Definition 2: The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using any percutaneous method. These measurements will be made by the independent angiographic core laboratory. If the core laboratory is unable to assess the % residual stenosis, the Investigator's assessment as recorded in the CRF will be used for the statistical analysis.
Procedure success | At the end of the index procedure or during hospital stay
  Definition 1: The attainment of <50% residual stenosis of the target lesion and no in-hospital MACE.
  Definition 2: The attainment of < 30% residual stenosis by QCA (or < 20% by visual assessment) AND a TIMI flow 3 after the procedure, using any percutaneous method without the occurrence of MACE during the hospital stay. These measurements will be made by the independent angiographic core laboratory. If the core laboratory is unable to assess the % residual stenosis, the Investigator's assessment as recorded in the CRF will be used for the statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Shuzheng Lv, Principal Investigator — An Zhen Hospital; Yundai Chen, Principal Investigator — Chinese PLA General Hospital; Zhimin Du, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University; Bo Xu, Principal Investigator — Beijing Fu Wai Hospital; Yuejin Yang, MD, Principal Investigator — Fu Wai Hospital, Beijing, China; Zuyi Yuan, Principal Investigator — First Affiliated Hospital of Medical College of ZI'AN Jiaotong University
Locations (4):
- China (4):
  - An Zhen Hospital, Beijing, Beijing Municipality
  - Beijing Fu Wai Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - First Affiliated Hospital of Medical College of XI'AN Jiaotong University, Xi'an, Shaanxi

REFERENCES:
- [Result] Xu B, Yang Y, Yuan Z, Du Z, Wong SC, Genereux P, Lu S; RESOLUTE China RCT Investigators. Zotarolimus- and paclitaxel-eluting stents in an all-comer population in China: the RESOLUTE China randomized controlled trial. JACC Cardiovasc Interv. 2013 Jul;6(7):664-70. doi: 10.1016/j.jcin.2013.03.001. Epub 2013 Mar 21. PMID 23523240